CLINICAL TRIAL: NCT01371032
Title: A Randomized, Prospective Study to Compare the Video Miller Device to Direct Laryngoscopy Using a Standard Pediatric Miller Blade for Tracheal Intubation of Children < 3 Years of Age Undergoing General Anesthesia
Brief Title: Study: Study to Compare Video Miller Device to Direct Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00024542
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Surgeries Undergoing General Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Miller laryngoscope (Active Comparator): using the screen (Video laryngoscopy group)
  Interventions: Device: VideoMiller
- Direct laryngoscopy (Active Comparator): without use the screen (Direct laryngoscopy group)
  Interventions: Device: Direct Laryngoscopy

INTERVENTIONS:
Device: VideoMiller — Video-Miller laryngoscope, using the screen (Video laryngoscopy group)
  Arms: Video-Miller laryngoscope
Device: Direct Laryngoscopy — Video-Miller laryngoscope, without screen (Direct laryngoscopy group)
  Arms: Direct laryngoscopy

SUMMARY:
The purpose of this study is to compare:

the standard pediatric intubation instrument (Miller blade) used as direct laryngoscopy during tracheal intubation to the VideoMiller device (the standard pediatric blade with a camera attached, giving indirect view of the vocal cords in the screen). This intubation device is used to place the tube in the trachea to keep the patient breathing during the surgery procedure.

The anesthesiologist obtains a better view of the vocal cords looking at the screen provided by the VideoMiller.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 3 years or younger undergoing anesthesia requiring endotracheal intubation.
2. Obtaining signed the informed consent by their parents or legal guardian.
3. American Society of Anaesthesiologists (ASA) physical status classification I - II or III

Exclusion Criteria:

1. Patients deemed to be at significant airway risk necessitating an awake fiber optic intubation
2. Patients with facial abnormalities, and/or oral-pharyngeal malformation.
3. Emergency operation

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD,PhD, Principal Investigator — Cedars-Sinai Medical Center; Ronald H Wender, MD, Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States

REFERENCES:
- [Derived] Lingappan K, Neveln N, Arnold JL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2023 May 12;5(5):CD009975. doi: 10.1002/14651858.CD009975.pub4. PMID 37171122

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.6 (4) | 9.6 (7) | 8 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 2 | 0 | 2
  Caucasian | 11 | 14 | 25
Weight [Mean (Standard Deviation); unit: Kg] | 8 (3) | 10 (4) | 9 (3)
Height [Mean (Standard Deviation); unit: cm] | 71 (13) | 69 (13) | 70 (13)
Laryngoscope Blade Size [Number; unit: Count of Participants] — Laryngoscope blades are used for examination of the interior of the larynx and for placement of an endotracheal tube. The Miller Laryngoscope Blades sizes (The most popular of the straight types) go from 0 to 4. For the pediatric ages used in this studies the sizes used were 0 and 1.
  Count of Participants
    Laryngoscope Blade size 0 | 12 | 13 | 25
    Laryngoscope Blade size 1 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Obtain Glottic View
Description: Time to obtain glottic view (from initial insertion of laryngoscope blade to obtain glottic view)
Time Frame: Times following initial insertion of laryngoscope blade to obtain glottic view
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Number analyzed (Participants) | 14 | 14
seconds | 9.2 (5) | 8.4 (6.4)

2. Primary Outcome: Intubation Time
Description: Times following initial insertion of laryngoscope blade to placement of tracheal tube
Time Frame: Times from insertion of laryngoscope blade to placement of tracheal tube
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Video-Miller Laryngoscope: Video-Miller laryngoscopy group (using the screen of the Video-Miller laryngoscope device for intubation)
- Direct Laryngoscopy: Direct laryngoscopy group (using the video-Miller laryngoscope, without access to the screen).
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Number analyzed (Participants) | 14 | 14
Seconds | 21 (11) | 28 (20)

3. Primary Outcome: Time From Insertion of Laryngoscope Blade to Confirm w/ CO2 Waveform
Description: Time following initial insertion of laryngoscope blade to confirm w/ CO2 waveform
Time Frame: Time from initial insertion of laryngoscope blade to confirm w/ CO2 waveform
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Number analyzed (Participants) | 14 | 14
seconds | 61 (37) | 59 (30)

4. Secondary Outcome: Glottis Visualization Using POGO Score
Description: POGO score represents the percentage of glottic opening seen (from 0-100%)
Time Frame: During intubation procedure, up to 3 minutes
Measure: Mean (Standard Deviation); unit: percentage of glottic opening
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Number analyzed (Participants) | 14 | 14
percentage of glottic opening | 94 (5.6) | 93.2 (14)

5. Secondary Outcome: Glottis Visualization Using Cormack Lehane
Description: Glottic visualization comparison between the two devices. Grade Description Approximate frequency Likelihood of difficult intubation
  1. Full view of glottis 68-74% <1%
  2. a Partial view of glottis 21-24% 4.3-13.4%
  2b Only posterior extremity of glottis seen or only arytenoid cartilages 3.3-6.5% 65-67.4% 3 Only epiglottis seen, none of glottis seen 1.2-1.6% 80-87.5% 4 Neither glottis nor epiglottis seen very rare
Time Frame: During intubation procedure, up to 3 minutes
Measure: Number; unit: Count of Participants
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Number analyzed (Participants) | 14 | 14
Count of Participants
  Cormack Lehane score 1 | 12 | 12
  Cormack Lehane score 2 | 2 | 2

6. Secondary Outcome: Number of Participants Intubated With 1 and > 1 Intubation Attempts
Description: Number of Participants intubated after 1 intubation attempt and Number of Participants intubated after > 1 intubation attempts
Time Frame: During intubation procedure, up to 3 minutes
Measure: Number; unit: participants
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
Number analyzed (Participants) | 14 | 14
participants
  Intubation attempt= 1 | 11 | 12
  Intubation attempts > 1 | 3 | 2

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Video-Miller Laryngoscope | Direct Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No